CLINICAL TRIAL: NCT00465582
Title: B14 Meningococcal Carriage in Seine-Maritime Population: Prevalence Study and Search of Risk Factors
Status: Terminated | Type: Observational
Sponsor: University Hospital, Rouen (Other)
Responsible Party: Sponsor
Other Study IDs: 2006/099/HP
Record Dates: First submitted 2007-04-24; First posted 2007-04-25 (Estimated); Last update posted 2012-03-27 (Estimated); Status verified 2012-03

CONDITIONS: Meningococcal Infections
Keywords: carriage; Neisseria meningitidis; risk factors
MeSH Terms: conditions — Meningococcal Infections

STUDY DESIGN:
Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — pharynx ecouvillonnage
Oversight: Data Monitoring Committee: Yes

SUMMARY:
Our main objectives are to evaluate the importance of meningococcal carriage and to determine the predisposing factors

ELIGIBILITY:
Inclusion Criteria:

* Living in the area of Dieppe
* Parental authority assent if necessary

Exclusion Criteria:

* Child under supervision

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Dieppe Population 0 to 25 yaers old.
Sampling Method: Non-Probability Sample
Enrollment: 3296 (Actual)
Dates: Start 2008-01; Study Completion 2008-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Francois Caron, Professor, Principal Investigator — Service des Maladies Infectieuses
Locations (1):
- François Caron, Rouen, Seine-Maritime, France